CLINICAL TRIAL: NCT01576263
Title: Autologous Blood Transfusion After Local Infiltration Analgesia With Ropivacaine in Total Knee and Hip Arthroplasty
Brief Title: Autologous Blood Transfusion After Local Infiltration
Status: Completed | Type: Observational
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: N-20090061
Record Dates: First submitted 2012-04-03; First posted 2012-04-12 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Total Hip Arthroplasty; Total Knee Arthroplasty
Keywords: Anaesthesia; Infiltration; Blood transfusion; Autologous; Arthroplasty; Replacement; Ropivacaine
MeSH Terms: interventions — Blood Transfusion, Autologous; Ropivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Venous blood to collect an analysis of total ropivacaine concentrations.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Total knee arthroplasty: 25 consecutive patients diagnosed for total knee arthroplasty.
  Interventions: Drug: Autologous blood transfusion with ropivacaine
- Total hip arthroplasty: 27 patients diagnosed for total hip arthroplasty.
  Interventions: Drug: Autologous blood transfusion with ropivacaine

INTERVENTIONS:
Drug: Autologous blood transfusion with ropivacaine — Local infiltration analgesia with ropivacaine 3 mg/kg, max 200 mg
  Other Names: No other names.
  Groups: Total knee arthroplasty
Drug: Autologous blood transfusion with ropivacaine — Local infiltration analgesia with ropivacaine 3 mg/kg, max 200 mg.
  Other Names: No other names.
  Groups: Total hip arthroplasty

SUMMARY:
Total knee and hip arthroplasty for osteoarthritis is performed on still broader indications even in elderly patients with previous or current medical conditions. Especially comorbidity like cardiovascular diseases and conditions with increased risk of bleeding or previous thrombo-embolic events are major challenges.

To facilitate safe use of ropivacaine as an analgesic, information on the concentrations levels after autologous blood transfusion following local infiltration analgesia is very crucial. However, very limited data are available. To verify the safety of autologous blood transfusion, ropivacaine concentrations were studied in 52 patients undergoing either total knee arthroplasty or total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis for hip arthroplasty
* Clinical diagnosis for knee arthroplasty

Exclusion Criteria:

* Patients < 18 years
* Lack of informed consent
* Inability to read/understand Danish
* Bilateral diagnosis
* Cancer diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2010-03; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Concentrations of ropivacaine in serum | 6 hours
  Concentrations of ropivacaine in serum before and after autologous blood transfusion will be analyzed.

SECONDARY OUTCOMES:
Analysis of ECG and pulse rate | 6 hours
  ECG, pulse rate and blood pressure will be analyzed in proportion to concentrations of serum before and after autologous blood transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Ole Simonsen, M.D., Principal Investigator — Northern Orthopaedic Department, Aalborg University Hospital, Denmark; Sten Rasmussen, M.D., Study Chair — Northern Orthopaedic Division, Aalborg University Hospital, Denmark; Bjarne B. Dencker, M.D., Study Chair — Department of Anaesthesiology, Aalborg University Hospital, Denmark; Torben Breindahl, M.D., Study Chair — Department of Clinical Biochemistry, Vendsyssel Hospital, Aarhus University, Denmark
Locations (1):
- Vendsyssel Hospital, Frederikshavn, Aalborg Hospital, Aarhus University, Aalborg, Denmark